CLINICAL TRIAL: NCT04002557
Title: Optimising Consultation Summaries to Promote Good Health/Views of Adolescents Attending Diabetes Clinic
Brief Title: Optimising Consultation Summaries to Promote Good Health
Acronym: ONSET
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4465
Record Dates: First submitted 2019-06-17; First posted 2019-06-28 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Type1 Diabetes
Keywords: diabetes; clinic letter; clinic summary; post-consultation letter
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus group: This is a qualitative study using focus group discussions with young people aged 12-18 who are receiving consultation summaries.
  Patients attending a single diabetes service will be invited to enrol. This service serves a population from a wide geographic area and socio-economic backgrounds.
  Interviews will be conducted by a qualitative researcher with relevant experience. They will be held on the day of a participant's clinic appointment within the same hospital or on the day agreed with the participant.
  Interventions: Other: Interview-Questionnaire

INTERVENTIONS:
Other: Interview-Questionnaire — Questionnaire

SUMMARY:
Patient participation in decision making about their care promotes patient satisfaction and confidence. Further more, allowing patients to see letters written about them enables trust, encourages patients to be involved in decision making process and allow patient understanding.

Little is known about how young people value these letters in the same way. Only one brief questionnaire study focused on adolescent views and found that young people wished to receive consultation summaries.

This research aims explore the views of adolescent patients related to consultation summaries that they receive following a doctor's appointment. The investigator will use patients attending a specialist diabetes clinic as our cohort and conduct a qualitative study using focus groups.

DETAILED DESCRIPTION:
Patient participation in decision making processes about their care promotes patient satisfaction and confidence. As part of this, allowing patients to see letters written about them enables trust, encourages patients to be involved in decision making process and allow patient understanding. Given this, the 2000 NHS plan made it a requirement that all medical correspondence between health professionals is shared with patients.

It is estimated that 40-80% of information discussed during a consultation is forgotten immediately. Written summaries have shown to be an effective method of improving patient recall of information by 20.8%.

The literature on the benefits/disadvantages of consultation summaries is largely focused on adult patients with little research done to explore the views of adolescent population. Where the patient is a child, the literature is only focussed on parents of children and not the children themselves. Limited research has shown that parents/care givers report clinic letters being useful in assisting with better understanding and management of their child's condition.

Little is known about how young people value these letters in the same way. Only one brief questionnaire study focused on adolescent views and found that young people wished to receive consultation summaries.

Adolescence is an important time of an individual's life. This is the time when many independent health behaviours are established. During adolescence, young people start showing more interest in their own health and often wish to participate in decision making processes regarding their care. The role of health workers at this stage is to appreciate young people as individuals . Clinic summaries addressed directly to young people might play an important role in assisting with establishment of health behaviours and promoting good health in young people.

The aim of this research is to understand the views of adolescent patients on consultation summaries and identify factors can improve these summaries and subsequently their health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years attending UCLH adolescent diabetes outpatient clinic

Exclusion Criteria:

* Young people who cannot speak English (effective communication with colleagues during the study is the major aspect of valid data collection)
* Young people who refuse to participate in focus group discussions

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Young people aged 12-18 years attending a single diabetes outpatient clinic were invited to enrol. This clinic served patients from a wide geographical area across London and the South-East England with broad socio-economic status, diabetes control and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Inwald, Principal Investigator — Imperial College London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bartle DG, Diskin L, Finlay F. Copies of clinic letters to the family. Arch Dis Child. 2004 Nov;89(11):1032-3. doi: 10.1136/adc.2004.051938. PMID 15499057
- [Background] Baxter S, Farrell K, Brown C, Clarke J, Davies H. Where have all the copy letters gone? A review of current practice in professional-patient correspondence. Patient Educ Couns. 2008 May;71(2):259-64. doi: 10.1016/j.pec.2007.12.002. Epub 2008 Jan 25. PMID 18222056
- [Background] Harris C, Boaden R. Copying letters to patients: the view of patients and health professionals. J Health Serv Res Policy. 2006 Jul;11(3):133-40. doi: 10.1258/135581906777641712. PMID 16824259
- [Background] Kessels RP. Patients' memory for medical information. J R Soc Med. 2003 May;96(5):219-22. doi: 10.1177/014107680309600504. No abstract available. PMID 12724430
- [Background] Chan Y, Irish JC, Wood SJ, Rotstein LE, Brown DH, Gullane PJ, Lockwood GA. Patient education and informed consent in head and neck surgery. Arch Otolaryngol Head Neck Surg. 2002 Nov;128(11):1269-74. doi: 10.1001/archotol.128.11.1269. PMID 12431168
- [Background] Lawton J, Waugh N, Noyes K, Barnard K, Harden J, Bath L, Stephen J, Rankin D. Improving communication and recall of information in paediatric diabetes consultations: a qualitative study of parents' experiences and views. BMC Pediatr. 2015 Jun 10;15:67. doi: 10.1186/s12887-015-0388-6. PMID 26054649
- [Background] Waterston T, San Lazaro C. Sending parents outpatient letters about their children: parents' and general practitioners' views. Qual Health Care. 1994 Sep;3(3):142-6. doi: 10.1136/qshc.3.3.142. PMID 10139411
- [Background] A new series starts: the ABC of adolescence. (2005). BMJ, 330(7486).
- See also: Good Practice Guidelines - Department of Health, 2004 — http://webarchive.nationalarchives.gov.uk/+/http://www.dh.gov.uk/en/Publicationsandstatistics/Publications/PublicationsPolicyAndGuidance/DH_4007561

RESULTS

PARTICIPANT FLOW:
Groups:
- Semi-structured Interview: This is a qualitative study using semi-structured interviews with young people aged 12-18 who are receiving consultation summaries.
  Patients attending a single diabetes service will be invited to enrol. This service serves a population from a wide geographic area and socio-economic backgrounds.
  Interviews will be conducted by a qualitative researcher with relevant experience. They will be held on the day of a participant's clinic appointment within the same hospital or on the day agreed with the participant.
  No intervention: Interviews contain no intervention, purely observational.
Period: Overall Study
Arm/Group | Semi-structured Interview
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Semi-Structured Interview
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants] — Participant's age was recorded
  Participants
    Age between 15 and 19 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Participant's gender was collected
  Participants
    Female | 5
    Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completed Interviews About Consultation Summaries They Were Receiving
Description: The aim of this research is to understand the views of adolescent patients on consultation summaries and identify factors can improve these summaries and subsequently their health and well-being.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Semi-structured Interview
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 month
Description: Semi-structure interview on a non-sensitive topic, risk of adverse events is minimal
Arm/Group | Semi-structured Interview
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-11-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT04002557/Prot_000.pdf